CLINICAL TRIAL: NCT00605917
Title: Special Investigation Of J Zoloft For Panic Disorder Patients
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0501092
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sertraline hydrochloride.: The patients of Panic disorder taking Sertraline hydrochloride.
  Interventions: Drug: Sertraline hydrochloride

INTERVENTIONS:
Drug: Sertraline hydrochloride — J ZOLOFT® Tablets 25 mg and J ZOLOFT® Tablets 50 mg. J ZOLOFT is Brand name in Japan.
  Dosage, Frequency: According to Japanese LPD, "The usual initial dose of J ZOLOFT in adults is 25 mg daily as sertraline and then gradually increased up to 100 mg, which should be given orally once daily. The dose may be adjusted within the range not exceeding 100mg according to the patient's age and symptoms".
  Duration: According to the protocol of A0501092, the duration of the investigation for findings regarding safety and efficacy of a panic disorder patient is from the first drug administration to the 16 weeks after the first administration.
  Other Names: J Zoloft, Zoloft

SUMMARY:
The objective of this surveillance is to collect information for panic disorder patients about 1) adverse drug reactions not expected from the LPD (unknown adverse drug reactions), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All patients with panic disorder to whom an investigator prescribes the first sertraline hydrochloride should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients with panic disorder need to be taking sertraline hydrochloride in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not taking sertraline hydrochloride.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients to whom an investigator involved in A0501092 prescribes sertraline hydrochloride.
Sampling Method: Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501092&StudyName=Special%20Investigation%20Of%20J%20Zoloft%20For%20Panic%20Disorder%20Patients%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert; This study is Special Investigation of JZOLOFT for panic disorder and one of conditions of this study is "patients who are diagnosed with panic disorder". So, all of participants in this study are panic disorder patients.
Period: Overall Study
Arm/Group | Sertraline
Started | 987
Completed | 908
Not Completed | 79
Not completed — Protocol Violation | 79

BASELINE CHARACTERISTICS:
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert
Arm/Group | Sertraline
Number analyzed (Participants) | 908
Age, Customized [Number; unit: participants]
  <65 years | 863
  >=65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 592
  Male | 316
Target Disease Severity [Number; unit: participants] — The severity of target disease which was diagnosed by investigator
  participants
    Mild | 325
    Moderate | 511
    Severe | 72
Complications [Number; unit: participants] — Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
  participants
    Present | 305
    Absent | 603
Concomitant drug [Number; unit: participants] — Concomitant drugs is the drugs which participant had taken during the observation period of this study to treat for participant's illnesses, injuries etc. The physician of this survey listed all of concomitant drugs. (e.g. paroxetine, milnacipran, etc.)
  participants
    Present | 671
    Absent | 237
Starting dose [Number; unit: participants] — Starting dose of each participant enrolled in this study
  participants
    25 mg | 699
    50 mg | 176
    75 mg | 18
    100 mg | 6
    other | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants of Treatment Related Adverse Events (TRAEs)
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: Baseline up to 52 weeks
Population: Safety analysis population included all enrolled participants who had received at least 1 confirmed administration of Sertraline.
Measure: Number; unit: participants
Groups:
- Sertraline: Participants who took Sertraline according to Japanese Package Insert
Arm/Group | Sertraline
Number analyzed (Participants) | 908
participants | 110

2. Primary Outcome: Number of Treatment Related Adverse Events (TRAEs) Not Expected From Japanese Package Insert
Time Frame: Baseline up to 52 weeks
Population: The safety analysis population consists of the cases that satisfy the participants conditions and in whom administration of Sertraline was confirmed.
Measure: Number; unit: events
Arm/Group | Sertraline
Number analyzed (Participants) | 908
events
  Sedation | 3
  Gastritis | 2
  Hyperuricaemia | 1
  Ventricular extrasystoles | 1

3. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Starting Dose
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether starting dose is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- 25mg: Participants whose starting dose were 25mg
- 50mg: Participants whose starting dose were 50mg
- 75mg: Participants whose starting dose were 75mg
- 100mg: Participants whose starting dose were 100mg
- Other Than Those Above: Participants whose starting dose were other than 25mg, 50mg, 75mg and 100mg
Arm/Group | 25mg | 50mg | 75mg | 100mg | Other Than Those Above
Number analyzed (Participants) | 699 | 176 | 18 | 6 | 9
participants | 101 | 6 | 0 | 0 | 3
Statistical Analysis 1: Comparison: 25mg vs 50mg vs 75mg vs 100mg vs Other Than Those Above; The risk factor tested was "starting dose". The null hypothesis is there is no difference between "three types of starting dose" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

4. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Concomitant Drug
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without concomitant drug is significant risk factor, Concomitant drugs is the drugs which participant had taken during the observation period of this study to treat for participant's illnesses, injuries etc. The physician of this survey listed all of concomitant drugs. (e.g. paroxetine, milnacipran, etc.)
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Concomitant Drug: Participants with concomitant drug who took Sertraline according to Japanese Package Insert
- Without Concomitant Drug: Participants without concomitant drug who took Sertraline according to Japanese Package Insert
Arm/Group | With Concomitant Drug | Without Concomitant Drug
Number analyzed (Participants) | 665 | 243
participants | 94 | 16
Statistical Analysis 1: Comparison: With Concomitant Drug vs Without Concomitant Drug; The risk factor tested was "concomitant drug". The null hypothesis is there is no difference between "with and without concomitant drug" in the participants of responders; Test type: Superiority or Other; p = 0.002, Chi-squared — not adjusted, p=0.050

5. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Family History of Psychiatric Disorder
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without family history of psychiatric disorder is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Family History: Participants with family history of psychiatric disorders who took Sertraline according to Japanese Package Insert
- Without Family History: Participants without family history of psychiatric disorders who took Sertraline according to Japanese Package Insert
Arm/Group | With Family History | Without Family History
Number analyzed (Participants) | 52 | 697
participants | 11 | 78
Statistical Analysis 1: Comparison: With Family History vs Without Family History; The risk factor tested was "family history of psychiatric disorder". The null hypothesis is there is no difference between "with and without family history of psychiatric disorder" in the participants of responders; Test type: Superiority or Other; p = 0.032, Chi-squared — not adjusted, p=0.050

6. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Smoking Status
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether smoking status is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Don't Smoke at All: Participants who didn't smoke at all and who took Sertraline according to Japanese Package Insert
- Used to Smoke But do Not Then: Participants who used to smoke but didn't then and who took Sertraline according to Japanese Package Insert
- Smoke Then: Participants who smoke then and who took Sertraline according to Japanese Package Insert
Arm/Group | Don't Smoke at All | Used to Smoke But do Not Then | Smoke Then
Number analyzed (Participants) | 542 | 31 | 142
participants | 57 | 9 | 30
Statistical Analysis 1: Comparison: Don't Smoke at All vs Used to Smoke But do Not Then vs Smoke Then; The risk factor tested was "smoking status". The null hypothesis is there is no difference between "three types of smoking status" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

7. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Past Medical History of Other Illness
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without past medical history of other illness is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Past Medical History of Other Illness: Participants with past medical history of other illness who took Sertraline according to Japanese Package Insert
- Without Past Medical History of Other Illness: Participants without past medical history of other illness who took Sertraline according to Japanese Package Insert
Arm/Group | With Past Medical History of Other Illness | Without Past Medical History of Other Illness
Number analyzed (Participants) | 103 | 805
participants | 25 | 85
Statistical Analysis 1: Comparison: With Past Medical History of Other Illness vs Without Past Medical History of Other Illness; The risk factor tested was "past medical history of other illness". The null hypothesis is there is no difference between "with and without past medical history of other illness" in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

8. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Non-Pharmaceutical Therapies
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without non-pharmaceutical therapies is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: The safety analysis population consists of the cases that satisfy the participants conditions and in whom administration of was confirmed.
Measure: Number; unit: participants
Groups:
- With Non-pharmaceutical Therapies: Participants with non-pharmaceutical therapies who took Sertraline according to Japanese Package Insert
- Without Non-pharmaceutical Therapies: Participants without non-pharmaceutical therapies who took Sertraline according to Japanese Package Insert
Arm/Group | With Non-pharmaceutical Therapies | Without Non-pharmaceutical Therapies
Number analyzed (Participants) | 405 | 503
participants | 65 | 45
Statistical Analysis 1: Comparison: With Non-pharmaceutical Therapies vs Without Non-pharmaceutical Therapies; The risk factor tested was "non-pharmaceutical therapies". The null hypothesis is there is no difference between "with and without non-pharmaceutical therapies" in the participants of responders; Test type: Superiority or Other; p = 0.001, Chi-squared — not adjusted, p=0.050

9. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: History of Treatment Prior to Administration of Sertraline
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without history of treatment prior to administration of Sertraline is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With History of Treatment: Participants with history of treatment prior to administration of Sertralin who took Sertraline according to Japanese Package Insert
- Without History of Treatment: Participants without history of treatment prior to administration of Sertralin who took Sertraline according to Japanese Package Insert
Arm/Group | With History of Treatment | Without History of Treatment
Number analyzed (Participants) | 200 | 679
participants | 33 | 73
Statistical Analysis 1: Comparison: With History of Treatment vs Without History of Treatment; The risk factor tested was "history of treatment prior to administration of Sertraline". The null hypothesis is there is no difference between "with and without history of treatment prior to administration of Sertraline" in the participants of responders; Test type: Superiority or Other; p = 0.028, Chi-squared — not adjusted, p=0.050

10. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Average Daily Dose
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without average daily dose is significant risk factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- <25mg: Participants who took less than 25mg of Sertraline a day on average according to Japanese Package Insert
- >=25mg, <50mg: Participants who took more than 25mg and less than 50mg of Sertraline a day on average according to Japanese Package Insert
- >=50mg, <75mg: Participants who took more than 50mg and less than 75mg of Sertraline a day on average according to Japanese Package Insert
- >=75mg, <100mg: Participants who took more than 75mg and less than 100mg of Sertraline a day on average according to Japanese Package Insert
- >=100mg: Participants who took more than 100mg of Sertraline a day on average according to Japanese Package Insert
Arm/Group | <25mg | >=25mg, <50mg | >=50mg, <75mg | >=75mg, <100mg | >=100mg
Number analyzed (Participants) | 13 | 529 | 211 | 151 | 4
participants | 2 | 92 | 14 | 2 | 0
Statistical Analysis 1: Comparison: <25mg vs >=25mg, <50mg vs >=50mg, <75mg vs >=75mg, <100mg vs >=100mg; The risk factor tested was "average daily dose". The null hypothesis is there is no difference of five types of average daily dose in the participants of responders; Test type: Superiority or Other; p < 0.001, Chi-squared — not adjusted, p=0.050

11. Secondary Outcome: Risk Factors for Incidence Rate of Treatment Related Adverse Events (TRAEs) of Sertraline: Complications
Description: Number of participants with Treatment Related Adverse Events (TRAEs) of Sertraline to determine whether with or without complications is significant risk factor, Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
Time Frame: Baseline up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- With Complications: Participants with complications who took Sertraline according to Japanese Package Insert
- Without Complications: Participants without complications who took Sertraline according to Japanese Package Insert
Arm/Group | With Complications | Without Complications
Number analyzed (Participants) | 305 | 603
participants | 47 | 63
Statistical Analysis 1: Comparison: With Complications vs Without Complications; The risk factor tested was "complications". The null hypothesis is there is no difference between "with and without complications" in the participants of responders; Test type: Superiority or Other; p = 0.030, Chi-squared — The risk factor tested was "complications". The null hypothesis is there is no difference between "with and without complications" in the participants of responders; not adjusted, p=0.050

12. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Concomitant Drug
Description: Number of participants with responders of Sertraline to determine whether with or without concomitant drug is significant factor
Time Frame: Baseline up to 52 weeks
Population: The efficacy analysis population consists of the evaluable cases in accordance with the analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Groups:
- Without Concomitrant: Participants without concomitant drug who took Sertraline according to Japanese Package Insert
Arm/Group | With Concomitant Drug | Without Concomitrant
Number analyzed (Participants) | 649 | 232
participants | 565 | 216
Statistical Analysis 1: Comparison: With Concomitant Drug vs Without Concomitrant; The factor tested was "concomitant drug". The null hypothesis is there is no difference between "with and without concomitant drug" in the participants of responders; Test type: Superiority or Other; p = 0.013, Chi-squared — not adjusted, p=0.050

13. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Complication
Description: Number of participants with responders of Sertraline to determine whether with or without complication is significant factor, Complications is the patient's current experiences with illnesses, operations, injuries and treatments. The physician of this survey made the diagnosis. (e.g. hypertension, diabetes, etc.)
Time Frame: Baseline up to 52 weeks
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | With Complications | Without Complications
Number analyzed (Participants) | 292 | 589
participants | 246 | 535
Statistical Analysis 1: Comparison: With Complications vs Without Complications; The factor tested was "complications". The null hypothesis is there is no difference between "with or without complications" in the participants of responders; Test type: Superiority or Other; p = 0.004, Chi-squared — not adjusted, p=0.050

14. Secondary Outcome: Factors Considered to Affect the Efficacy of Sertraline: Drinking Status
Description: Number of participants with responders of Sertraline to determine whether drinking status is significant factor
Time Frame: Baseline up to 52 weeks
Population: as for outcome 12
Measure: Number; unit: participants
Groups:
- Didn't Drink Alcohol at All, and Had Never Drunk Alcohol: Participants who didn't drink alcohol at all, and had never drunk alcohol and who took Sertraline according to Japanese Package Insert
- Drank Alcohol Very Occasionally: Participants who drank alcohol very occasionally and who took Sertraline according to Japanese Package Insert
- Used to Drink Alcohol But Did Not Then: Participants who used to drink alcohol but did not then and who took Sertraline according to Japanese Package Insert
- Drank Alcohol Moderately: Participants who drank alcohol moderately and who took Sertraline according to Japanese Package Insert
- Drank Alcohol Every Day: Participants who drank alcohol every day and who took Sertraline according to Japanese Package Insert
Arm/Group | Didn't Drink Alcohol at All, and Had Never Drunk Alcohol | Drank Alcohol Very Occasionally | Used to Drink Alcohol But Did Not Then | Drank Alcohol Moderately | Drank Alcohol Every Day
Number analyzed (Participants) | 200 | 335 | 28 | 128 | 65
participants | 171 | 312 | 23 | 118 | 53
Statistical Analysis 1: Comparison: Didn't Drink Alcohol at All, and Had Never Drunk Alcohol vs Drank Alcohol Very Occasionally vs Used to Drink Alcohol But Did Not Then vs Drank Alcohol Moderately vs Drank Alcohol Every Day; The factor tested was "drinking status". The null hypothesis is there is no difference between "five types of drinking status" in the participants of responders; Test type: Superiority or Other; p = 0.004, Chi-squared — not adjusted, p=0.050

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Sertraline: Participants taking Sertraline according to Japanese Package Insert.The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Arm/Group | Sertraline
Serious Adverse Events (participants affected / at risk) | 1/908
Other Adverse Events (participants affected / at risk) | 110/908
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=908)
Mania (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=908)
Nausea (Gastrointestinal disorders) | 31 (31)
Somnolence (Nervous system disorders) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 13 (13)
Abdominal discomfort (Gastrointestinal disorders) | 9 (9)
Headache (Nervous system disorders) | 6 (6)
Malaise (General disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Sedation (Nervous system disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Terminal insomnia (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1)
Ejaculation failure (Reproductive system and breast disorders) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.